CLINICAL TRIAL: NCT05683899
Title: Evaluation of Emergency Department AI Prediction Algorithm
Brief Title: A Study of Emergency Department AI Prediction Impact
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Alexander J. Ryu, Principal Investigator, Mayo Clinic
Other Study IDs: 22-011319
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Hospital Admission; Length of Stay
Keywords: AI Prediction Algorithm; Emergency Department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: 141 days with AI scores displayed
- Group B: 141 days with AI scores not displayed

SUMMARY:
The purpose of this study is to evaluate the impact of an AI admission prediction tool on the number of preventable hospital admissions, emergency department (ED) length of stay, when the predictions are displayed only to a dedicated ED triage team. Also, to evaluate user perceptions of the AI tool among the triage team users and medical officer of the day users. Additionally, to evaluate any impact of the AI tool on the number of interventions performed by the triage team, and to evaluate the impact of the tool on time-to-admission after an admission order is placed.

ELIGIBILITY:
Inclusion Criteria:

* For the survey component, any HIM clinician that works a shift in the triage area, ED physicians, and the medical officer of the day will be included.
* For length of stay data, adult patients registered in the Mayo Clinic-Rochester St. Mary's Emergency Department will be included.

Exclusion Criteria:

* For the survey, clinicians not working a triage shift during the study period will be excluded.
* For the length of stay analysis, only adult ED patients will be included, who do not triaged to the behavioral health/psychiatry pathway, nor patients who are triaged to the Emergency Department observation pathway.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The group being surveyed will consist of Hospital Internal Medicine (HIM) clinicians, (physicians, nurse practioners, and physician assistants) at the Mayo Clinic- Rochester site, who are all adults. The patients which are triaged by this group are only adults, and accordingly, the AI score will never be shown for pediatric patients, or patients undergoing psychiatric evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Hospital Admissions | 282 days
  Number of avoidable admissions prevented as a fraction of all ED patients in a day, specifically, the number of patients who were seen by the SAPPHIRE triage team and discharged home

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Ryu, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials